CLINICAL TRIAL: NCT01349218
Title: In Infants and Newborns, is There a Relation Between the Potassium Level in Blood Samples Drawn From a Vein and Those Drawn From a Heel Stick?
Brief Title: Relationship Between Potassium Level in Venous Blood Samples Drawn and Heel Sticks In Infants and Newborns
Acronym: PS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Memorial Hermann Hospital (Other)
Responsible Party: Principal Investigator, Samia Khalil, Professor - Anesthesiology, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HSC-MS-10-0180
Record Dates: First submitted 2011-05-03; First posted 2011-05-06 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Hyperkalemia
Keywords: Potassium; Infants; Heel Stick; Less than or equal to 6 months of age; IV catheter blood samples; perioperatively; elective surgical procedures
MeSH Terms: conditions — Hyperkalemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Blood sample drawn from a vein and from a heel stick (Experimental): 0.5 ml will be drawn from a vein when an IV is started for the surgery or from an IV already in place. The blood will be placed into a heparinized, 1 ml syringe for venous blood gas analysis. A second blood sample, 0.3 ml will be drawn into a capillary pipette from a heel stick for capillary blood gas analysis.
  Interventions: Other: Blood sample drawn from a vein; Other: Blood sample drawn from a heel stick

INTERVENTIONS:
Other: Blood sample drawn from a vein — 0.5 ml will be drawn from a vein when an IV is started for the surgery or from an IV already in place. The blood will be placed into a heparinized, 1 ml syringe for venous blood gas analysis.
Other: Blood sample drawn from a heel stick — A second blood sample, 0.3 ml will be drawn into a capillary pipette from a heel stick for capillary blood gas analysis.

SUMMARY:
The purpose of this study is to find out whether there is a correlation (link) between the level of potassium in blood samples drawn from a vein and those drawn from a heel stick in infants scheduled for elective surgery.

DETAILED DESCRIPTION:
This is a prospective study which will take place at the Children's Memorial Hermann Hospital Operating Room.

After obtaining written informed consent from parents or guardians, infants and babies scheduled to have elective surgery under routine general anesthesia and are <6 months of age will be included in the study. After the baby receives routine general anesthesia, a small amount of blood, 0.5 ml, will be drawn from a vein when an I.V. is started for the surgery. The largest possible cannula will be placed whenever possible to decrease hemolysis. If a baby has a central line, the blood sample will be drawn from it. If a baby has an existing peripheral I.V., a blood sample will be drawn from the I.V. cannula only if blood is freely running, to avoid hemolysis.

Blood will be placed into a heparinized, 1 ml syringe for venous blood gas analysis. A second blood sample, 0.3 ml, will be drawn into a capillary pipette from a heel stick for capillary blood gas analysis. The heel will be properly sterilized, and a proper size lancet will be used. The same operator will be performing the heel stick in each case.

ELIGIBILITY:
Inclusion Criteria:

* Infants and babies, ASA physical Status I-III, less than 6 month of age and scheduled to have elective surgery under routine general anesthesia at Children's Memorial Hermann Hospital will be included.

Exclusion Criteria:

* Babies and infants with documented anemia (< 8 gm), who are bleeding, ASA Classification >III, have sickle cell disease or trait, thalassemia, HIV or DIC will be excluded from the study. Babies with organ failure will be excluded.

Max Age: 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 31 (Actual)
Dates: Start 2014-03; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
Potassium Measurements | 0-30 minutes after start of surgery
  In this prospective study, we would like to evaluate whether there is a correlation between the potassium level in blood samples drawn from a vein and those drawn from a heel stick.

CONTACTS AND LOCATIONS:
Overall Officials: Samia N Khalil, M.D., Principal Investigator — Faculty
Locations (1):
- Memorial Hermann Hospital, Houston, Texas, United States